CLINICAL TRIAL: NCT06162819
Title: Efficacy of Flunarizine Vs Amitriptyline in Prophylaxis of Migraine Prophylaxis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shalamar Institute of Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: R&ID003
Record Dates: First submitted 2023-11-30; First posted 2023-12-08 (Actual); Last update posted 2023-12-29 (Actual); Status verified 2023-12

CONDITIONS: Migraine; Prophylaxis
MeSH Terms: conditions — Migraine Disorders | interventions — Amitriptyline; Flunarizine

STUDY DESIGN:
Intervention Model Description: Single blind, Randomized Parallel study design, All the consented participants will be randomized into two equal groups
Who Masked: Participant
Masking Description: Patients with migraine with even No. Medical Record will be assigned Amitriptyline whereas subjects with Odd Medical record No. will be treated with Flunarizine
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GroupA (Experimental): Amitriptyline group will be assessed at baseline and will be followed up at 6th week after treatment and at 12th week after treatment
  Interventions: Drug: Amitriptyline
- Group B (Experimental): Flunarizine group will be assessed at baseline and will be followed up at 6th week after treatment and at 12th week after treatment
  Interventions: Drug: Flunarizine 5mg

INTERVENTIONS:
Drug: Amitriptyline — Amitriptyline will be used for prophylaxis of migraine, also used as antidepressant
  Other Names: Amyline
  Arms: GroupA
Drug: Flunarizine 5mg — Flunarizine will be used for prophylaxis of migraine,
  Other Names: Sibelium
  Arms: Group B

SUMMARY:
To compare the frequency of acute attack and mean pain score ( assessed by visual analog scale) among subjects using either flunarizine or amitriptyline among patients with migraine coming to tertiary care Hospital in Lahore, Pakistan.

In this study 84 patients with migraine Age ranged between 18- 60 years, Both genders having 3 or more migraine attacks per month, normal systemic and neurological examination and not having taken any prophylactic medication for the last 4 months will randomly divided into two equal group of 42 subjects each.

DETAILED DESCRIPTION:
Introduction:

Migraine is a genetically influenced complex disorder characterized by episodes of moderate-to-severe headache, most often unilateral and generally associated with nausea and increased sensitivity to light and sound. Migraine is a common cause of disability and loss of work. Migraine attacks are complex brain events that unfold over hours to days in a recurrent matter. Migraine can be classified into subtypes according to the headache classification committee of the International Headache Society these subtypes include migraine without aura, migraine with aura and chronic migraine. Etiology of migraine in related to genetic, dietary and environmental factors. Acute migraine attack is characterized in to four phases of prodrome, aura headache and postdrome. Migraine has an approximate prevalence of 14.7% globally, making it the third most common disease in the world. It occurs three times more commonly in women as compared to men, which is most probably due to hormonal differences. The migraine attacks were most frequently triggered by sleep disturbance (70.5%), stress (66.7%), fatigue (64.4%), excess screen time (61.1%), loud noise (58.8%), dehydration (49.9%), and missed meals or dieting (49.1%). Other common triggering factors were traveling (39.9%), bright sunshine (39.2%), and certain smells or perfume (30.8%). The migraine attacks were triggered by smoking in only 8.1% of the migraineurs and by exercise in only 10.4% of the migraineurs.4 The global prevalence of migraine has increased substantially over the last three decades. According to the Global Burden of Disease (GBD) 2019 study, the estimated global prevalence of migraine increased from 721.9 million in 1990 to 1.1 billion in 2019. Treatment of migraine is divided into abortive measures for an acute attack and prophylactic measures to decrease frequency, severity and duration of attacks. Acute treatment aims to stop the progression of a headache quickly and therapy consists of stratified options of pharmacological and non-pharmacological measures, these include non-steroidal anti-inflammatory drugs, triptans, ergot derivate, dexamethasonse, Transcutaneous electrical nerve stimulation (TENS) therapy and occipital nerve block.

Recent studies have emphasized the role of prophylactic treatment of migraine because once an acute attack occurs, it often incapacitating its sufferers, reduce quality of life and cause significant disability. Preventive treatment aims to reduce attack frequency, improve responsiveness to acute attacks severity and duration, and reduce disability. Indications for preventive treatment include but not limited to frequent or long-lasting headaches, failure of acute therapy, and migraine with complications. Preventive treatment agents include beta blockers e.g. metoprolol and propranolol - especially in hypertensive and non-smoker patients, anti-depressants, amitriptyline and venlafaxine - especially in patients with depression or anxiety disorders and insomnia, Anticonvulsants: valproate acid and topiramate - especially in epileptic patients and Calcitonin gene-related peptide antagonists: erenumab, fremanezumab, and galcanezumab. Along with pharmacological measures life style changes must be a commitment from patient and these include regular exercise, avoidance of dietary triggers and cognitive-behavioural therapy

ELIGIBILITY:
Inclusion Criteria:

* Age 18- 60 years 2. Both genders 3. 3 or more migraine attacks per month 4. normal systemic and neurological examination 5. not having taken any prophylactic medication for the last 4 months

Exclusion Criteria:

* Un controlled hypertension 2. Ischemic heart disease, chronic liver failure and chronic liver disease 3. Pregnant patient 4. Known allergies to drug being used in study 5. Major pathology or surgery at the neck or the head 6. Recent injury or road traffic injury at the head or the cervical spine 7. Cancer pain 8. Rheumatological or immune related diseases 9. Implantable metallic or electrical devices in the head 10. Patients using opioids or user of illicit drugs or has had recent history of alcohol or drug abuse.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 84 (Estimated)
Dates: Start 2024-01-01 (Estimated); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
Severity of headache | It will be asses at baseline, at 6th week, and at 12th week
  pain severity will be assessed using Visual Analogue Scale (VAS)
No. of Attacks per month | It will be asses at baseline, at 6th week, and at 12th week
  reduction in number of attacks

CONTACTS AND LOCATIONS:
Overall Officials: Mujeeb-ur-Rehman Abid Butt, FCPS, Study Director — Shalamar Institute of Health Sciences
Locations (1):
- Shalamar Hospital, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No
Over all results will be presented in the form of publication.

REFERENCES:
- [Background] Gorur K, Gur H, Ismi O, Ozcan C, Vayisoglu Y. The effectiveness of propranolol, flunarizine, amitriptyline and botulinum toxin in vestibular migraine complaints and prophylaxis: a non-randomized controlled study. Braz J Otorhinolaryngol. 2022 Nov-Dec;88(6):975-981. doi: 10.1016/j.bjorl.2021.02.005. Epub 2021 Mar 7. PMID 33722518
- [Result] Athar F, Zahid A, Farooq M, Ayyan M, Ashraf M, Farooq M, Naeem F, Badar A, Ehsan M, Hussain A, Ilyas MA. Frequency of migraine according to the ICHD-3 criteria and its association with sociodemographic and triggering factors in Pakistan: A cross-sectional study. Ann Med Surg (Lond). 2022 Sep 17;82:104589. doi: 10.1016/j.amsu.2022.104589. eCollection 2022 Oct. PMID 36268304
- [Result] Amiri P, Kazeminasab S, Nejadghaderi SA, Mohammadinasab R, Pourfathi H, Araj-Khodaei M, Sullman MJM, Kolahi AA, Safiri S. Migraine: A Review on Its History, Global Epidemiology, Risk Factors, and Comorbidities. Front Neurol. 2022 Feb 23;12:800605. doi: 10.3389/fneur.2021.800605. eCollection 2021. PMID 35281991
- [Result] Bendtsen L, Sacco S, Ashina M, Mitsikostas D, Ahmed F, Pozo-Rosich P, Martelletti P. Guideline on the use of onabotulinumtoxinA in chronic migraine: a consensus statement from the European Headache Federation. J Headache Pain. 2018 Sep 26;19(1):91. doi: 10.1186/s10194-018-0921-8. PMID 30259200